CLINICAL TRIAL: NCT06375434
Title: The Mechanistic Study on the Influence of Gut Microbiota on Radiotherapy Sensitivity in Patients With Locally Advanced Rectal Cancer
Brief Title: Correlation Between Gut Microbiota and Radiosensitivity of Rectal Cancer
Acronym: GMRSC-LARC
Status: Not yet recruiting | Type: Observational
Sponsor: Jing-kun Liu (Other)
Responsible Party: Sponsor-Investigator, Jing-kun Liu, Principal Investigator, Xinjiang Medical University
Organization: Xinjiang Medical University (Other)
Other Study IDs: 20240101-01
Record Dates: First submitted 2024-04-12; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Locally Advanced Rectal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Feces；Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radiosensitive group
  Interventions: Other: No intervention
- The radiotherapy-insensitive group
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this process is to clarify the characteristics of gut microbiota changes in patients with locally advanced rectal cancer undergoing preoperative neoadjuvant treatment, and to identify key bacterial species closely related to sensitivity to radiotherapy. This aims to elucidate the mechanism linking gut microbiome dysbiosis with radiotherapy sensitivity, thereby providing new combined treatment strategies to enhance the efficacy of radiotherapy.

DETAILED DESCRIPTION:
The study is expected to enroll 100 patients with locally advanced rectal cancer, including 50 patients in the radiotherapy-sensitive group and 50 in the radiotherapy-resistant group. Each participant will provide stool and blood samples before treatment for subsequent metagenomic and metabolomic sequencing analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with late-stage rectal cancer (stages IIIB to IV), including those with postoperative recurrence re-staging or those intending to receive neoadjuvant treatment,
2. Pathological type is adenocarcinoma,
3. Have measurable lesions before radiotherapy or chemotherapy,
4. Age between 18 and 75 years,
5. A WHO Performance Status (PS) score of 0 to 2, capable of tolerating radiotherapy or chemotherapy,
6. An expected survival period of 6 months or more;
7. Able to understand the study and sign the informed consent form.

Exclusion Criteria:

1. Patients with severe complications or other malignant diseases.
2. Known severe allergic reactions to components of radiotherapy or chemotherapy.
3. Significant cardiac, hepatic, renal, or other vital organ dysfunction.
4. Pregnant or breastfeeding women.
5. Patients unable to comply with study requirements or affected by psychiatric or psychological diseases.
6. Participation in other clinical trials recently that could affect the assessment of this study's results.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will enroll 100 patients with locally advanced rectal cancer, aged 18-75, scheduled for neoadjuvant treatment. Participants will be divided into two groups of 50: one sensitive to radiotherapy and the other resistant. Each will provide stool and blood samples for metagenomic and metabolomic sequencing to investigate the gut microbiome's role in radiotherapy sensitivity. This will aid in identifying predictive biomarkers for personalized treatment strategies.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Diameter of tumor | 30 days
  The tumor diameter before and after radiotherapy and the reduced tumor diameter after treatment were calculated

SECONDARY OUTCOMES:
Change in Gut Microbiota Composition | 30 days
  Change in gut microbiota composition, including alterations in bacterial taxa, diversity, and abundance, between rectal cancer patients sensitive to radiotherapy and a control group of patients insensitive to radiotherapy.
Change in Plasma metabolites | 30 days
  Metabolomics sequencing, including profiling of metabolites and their differences, was performed on patients' plasma before radiotherapy.

OTHER OUTCOMES:
Five-year survival rate | 5 year